CLINICAL TRIAL: NCT00568789
Title: A Study of the Safety of Ramelteon in Elderly Subjects
Brief Title: Safety of Ramelteon in Elderly Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-375-060; U1111-1115-1906 (Registry Identifier: WHO)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia
Keywords: Insomnia; Aged; Postural Balance; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramelteon 8 mg, zolpidem 10 mg and placebo (Experimental)
  Interventions: Drug: Ramelteon, zolpidem and placebo

INTERVENTIONS:
Drug: Ramelteon, zolpidem and placebo — Ramelteon 8 mg, tablets, orally, one night only during Period 1, 2 or 3
  Zolpidem 10 mg, tablets, orally, one night only during Period 1, 2 or 3
  Ramelteon/Zolpidem placebo-matching tablets, orally one night only during Period 1, 2 or 3
  Other Names: Ambien; Rozerem™; TAK-375; ramelteon

SUMMARY:
The purpose of this study is to investigate the effects of ramelteon in elderly subjects on balance, mobility and memory impairment after awakening in the middle of the night following bedtime dosing.

DETAILED DESCRIPTION:
Insomnia affects more than half of the US population. Epidemiological data indicate that between 36% and 56% of American adults report occasional insomnia, while 9% to 17% report chronic or severe problems with insomnia. This condition is most prevalent in the elderly. Elderly insomnia sufferers may experience more difficulty staying asleep than younger adults; increasing wakefulness during the sleep period and resulting in the opportunity to get out of bed.

Elderly individuals with insomnia are at risk of falling when they get out of bed during the sleep period. It is not known if this risk merely is the result of being out of bed, or if insomnia or some other physiological processes (eg, postural hypotension) contribute. This risk is significant because falling may result in severe injuries, including hip fractures, for which morbidity and mortality statistics are remarkable. Approximately one-third of those who sustain a hip fracture are placed in long-term care facilities. Of those patients hospitalized due to a hip fracture, 15% die while in the hospital and 33% die within one year of sustaining the fracture.

One important concern regarding the risk of falling in elderly patients with insomnia relates to the commonly accepted pharmacological treatments of insomnia. Although normal control of the sleep-wake cycle is exerted by the suprachiasmatic nucleus via melatonin receptor subtypes 1 and 2 receptors, current pharmacologic treatments for insomnia mainly involve GABAergic (gamma aminobutyric acid) mechanisms: most currently prescribed sleep agents are benzodiazepine receptor agonists, which bind to the benzodiazepine receptor site of the gamma aminobutyric acid receptor complex. Gamma aminobutyric acid is the major inhibitory transmitter in the central nervous system and its receptors are distributed widely throughout the brain. In addition to sleep, benzodiazepine receptor agonists can cause a wide range of ancillary effects not directly related to sleep, depending on the precise subset of gamma aminobutyric acid receptors activated. These include sedative, anxiolytic, muscle-relaxant, and amnesic effects. Drugs that act at this receptor complex, specifically the benzodiazepines, have deleterious effects on body sway.

Ramelteon is marketed in the United States as Rozerem for the treatment of insomnia characterized by difficulty with sleep initiation. It's mechanism of action is based on the agonism of melatonin receptor subtype 1 and 2.

This study will investigate the effects of ramelteon on balance, mobility and memory impairment awakening in the middle of the night following bedtime dosing. Participation in this study is anticipated to be about 1 to 1.5 months.

ELIGIBILITY:
Inclusion Criteria

* Self-reported sleep latency of 30 minutes or greater on at least 3 nights per week during the last 3 months.
* Body mass index between 18 and 34, inclusive
* Habitual bedtime between 9 pm and 1 am.

Exclusion Criteria

* Performance outside of normal limits on the EquiTest Motor Control Test at the Screening Visit.
* Average score on the EquiTest Sensory Organization Test #5 of less than 40 at the Screening Visit.
* Average score on the EquiTest Sensory Organization Test #6 of less than 40 at the Screening Visit.
* History of sleep apnea, restless leg syndrome, period limb movement syndrome, or other known disorders which affect sleep with the exception of insomnia.
* Current vestibular system disorder or inner ear disease.
* Recent history of clinically significant head injury.
* Significant visual acuity or field abnormalities that are not improved with the use of corrective lenses.
* History of balance disturbance or frequent falling.
* History of seizures, strokes, degenerative neurological disease, fibromyalgia, diabetic neuropathy, thyroid dysfunction, hypotension, clinically significant arthritis or musculoskeletal disorder.
* History of cancer, other than basal cell carcinoma, that has not been in remission for at least five years prior to the first dose of study drug.
* Current significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable.
* Acute clinically significant illness within two weeks or has been hospitalized within four weeks prior to the Screening Visit.
* History of treatment for a psychiatric disorder (including anxiety, depression, mental retardation, cognitive disorder, bipolar illness and schizophrenia) within the past six months.
* History of drug addiction or drug abuse within the past 12 months, as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised.
* History of alcohol abuse within the past 12 months.
* Any clinically important abnormal finding, as determined by medical history, physical examination, electrocardiogram or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel.
* Positive urine drug screen for drugs known to alter sleep.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to the first dose of single-blind study medication, whichever is longer.
* Any additional condition that in the Investigator's opinion would:

  * affect sleep-wake function
  * prohibit the subject from completing the study
  * not be in the best interest of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Melatonin and all other drugs or supplements known to affect sleep/wake function
  * Anxiolytics
  * Sedatives
  * Hypnotics
  * Central nervous system active drugs (including herbal)
  * Antidepressants
  * Narcotic analgesics
  * Anticonvulsants
  * Beta blockers
  * Sedating H1 antihistamines
  * St. John's Wort
  * Systemic steroids
  * Kava-kava
  * Respiratory stimulants
  * Ginkgo-biloba
  * Decongestants
  * Over-the-counter and prescription stimulants
  * Antipsychotics
  * Over-the-counter and prescription diet aids
  * Muscle relaxants

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Sensory Organization Test Composite Score. | Periods 1, 2, and 3 in the evening before sleep and during night when awakened from sleep.

SECONDARY OUTCOMES:
Equilibrium Score (ES) for SOT conditions 5 and 6 (evaluation of the effect of ramelteon on balance). | Periods 1, 2, and 3 during night when awakened from sleep and in the morning after self-awakening.
Sensory Organization Test derived ratios: Somatosensory, Visual, Vestibular, and Preference (effect on balance). | Periods 1, 2, and 3 in the evening before sleep and during night when awakened from sleep.
Results of the Step/Quick Turn Test (SQTT), which quantifies turn performance characteristics, were obtained with NeuroCom EquiTest computerized dynamic posturography equipment (effect on mobility and balance). | Periods 1, 2, and 3 during night when awakened from sleep and in the morning after self-awakening.
Immediate Memory Recall Test. | Periods 1, 2, and 3 during night when awakened from sleep.
Delayed Recall Test. | Periods 1, 2, and 3 during night when awakened from sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (6):
- United States (6):
  - Costa Mesa, California
  - San Diego, California
  - Miami, Florida
  - Miramar, Florida
  - Orlando, Florida
  - New York, New York

REFERENCES:
- [Result] Zammit G, Wang-Weigand S, Peng X. Use of computerized dynamic posturography to assess balance in older adults after nighttime awakenings using zolpidem as a reference. BMC Geriatr. 2008 Jul 15;8:15. doi: 10.1186/1471-2318-8-15. PMID 18627623
- [Result] Zammit G, Wang-Weigand S, Rosenthal M, Peng X. Effect of ramelteon on middle-of-the-night balance in older adults with chronic insomnia. J Clin Sleep Med. 2009 Feb 15;5(1):34-40. PMID 19317379
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI